CLINICAL TRIAL: NCT01457599
Title: Computertomography-guided Wire Marking of Colorectal Hepatic Metastases After Complete Response to Neoadjuvant Chemotherapy. A Pilot Study
Brief Title: Computertomography-guided Wire Marking of the Liver
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Kornprat Peter, MD, MD, Medical University of Graz
Other Study IDs: INS-621000-0274-002
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Secondary Malignant Neoplasm of Liver
Keywords: liver-colorectal metastases-computertomography-guided-wire-chemotherapy-complete response; Feasibility, safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Marking Liver
  Interventions: Procedure: Computertomography-guided marking of colorectal liver metastases

INTERVENTIONS:
Procedure: Computertomography-guided marking of colorectal liver metastases — Computertomography-guided marking of colorectal liver metastases

SUMMARY:
The aim of the study is to evaluate if it is possible to mark with a wire colorectal hepatic metastases after complete response to a neoadjuvant chemotherapy.Primary the investigators want to investigate if the wire marking is a possibility to mark respectively to identify these lesions. Further the investigators want to evaluate how many patients with complete radiologic have complete histologic response in their specimen respectively in how many specimens in the definitive histology tumor cells are visible.

DETAILED DESCRIPTION:
Colorectal Cancer is most common in western countries. In 2007 in Austria 4462 new colorectal cancers were diagnosed. The most common place of metastasis is the liver. Approximately 15% of patients have metastasis at time of diagnosis of primary tumor and further 50% will develop metastases in the further course of the disease.However only 10-25% of patients are candidates for liver resection. New chemotherapeutics, new targeted therapies with monoclonal antibodies and better surgical techniques improved response rates, resection rates and overall survival. Owing to improved response rates metastases in the liver partially respectively completely disappeared, so that these lesions are not more visible in apparative diagnostic like CT-scan and MRI.

The question is now what to do with this patients? In the literature there is no evidence how to manage these patients. Conservative management would lead to a reoccurrence of metastases in the liver. On the other side surgical management is difficult, because metastases are preoperatively and intraoperatively not visible and resection is only possible with the removement of greater amounts of healthy tissue.

The computer tomography-guided wire marking of the metastases in the liver is a possibility to overcome these problems. All patients with complete radiologic response of metastases in the liver and metastases ≤ 1 cm are included in the study (RECISTE-Criteria). On day of surgical procedure patients will brought to interventional radiologist and based on computer tomography images before neoadjuvant chemotherapy the lesions will be marked computer tomography-guided with a wire(X-Reidy Breast Lesion Localization Needle, Cook Medical). The wire is placed percutaneously and under antibiotic prophylaxis. After the marking procedure, the patient is brought into the operating room to resect the metastases in the liver.

ELIGIBILITY:
Inclusion Criteria:

* Histologic verified cancer of the colon and rectum with metastases into the liver
* Neoadjuvant chemotherapy with complete radiologic response of metastases in apparative diagnostic respectively metastases with a diameter ≤ 1 cm.
* Technically Resectability
* Age ≥ 18 Years
* Written informed consent

Exclusion Criteria:

* Age < 18 Years
* Technically Irresectability
* Neoadjuvant chemotherapy and response of metastases, however with a diameter > 1 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity | One Year
  Sensitivity of wire marking to find liver metastases with complete response to neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided